CLINICAL TRIAL: NCT03684733
Title: Magnetic Resonance Breast Tissue Characterisation to Improve Risk Stratification for Breast Cancer
Acronym: MR-BTC
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 4173
Record Dates: First submitted 2018-04-27; First posted 2018-09-26 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation; Mammography; MRI
Keywords: Breast cancer; BRCA1/2 mutation carriers; Breast screening; Magnetic Resonance Imaging (MRI); X-ray mammography (XRM); Background Parenchymal Enhancement (BPE)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Arm 1: Cohort 1 - Retrospective Analysis: Participants attending MRI & XRM for a clinical indication with at least one normal breast
  Interventions: Diagnostic Test: MRI
- Arm 2: Cohort 2 - Retrospective Analysis: BRCA1 or BRCA2 mutation carriers attending MRI & XRM for breast screening:
  Genetic risk of breast cancer
  Interventions: Diagnostic Test: MRI
- Arm 2: Cohort 3 - Retrospective Analysis: Participants attending MRI & XRM for breast screening post mantle radiotherapy:
  Environmental risk of breast cancer
  Interventions: Diagnostic Test: MRI
- Arm 2: Cohort 4 - Prospective: General population attending XRM for breast investigation:
  Population risk of breast cancer MRI
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Clinical MRI breast screening examination

SUMMARY:
This is a combination retrospective/prospective observational study with two arms:

DETAILED DESCRIPTION:
Arm 1 :To establish the accuracy of MRI measurements from clinical MRI sequences

Cohort 1: Participants attending MRI & XRM for a clinical indication with at least one normal breast

Women attend MRI and XRM at the Royal Marsden NHS Foundation Trust for a wide range of clinical indications, including screening, staging and disease monitoring. Investigators will retrospectively analyse MRI and XRM examinations from women with at least one normal breast. This will enable a comparison of clinical and research MRI techniques to measure MRI Breast Density and BPE together with a correlation against PMD. This cohort should cover a wide range of ages and breast densities which will enable a useful comparison of measurement techniques.

Arm 2 To compare breast tissue between women at varying risk of breast cancer

Cohort 2: BRCA1 or BRCA2 mutation carriers attending MRI & XRM for breast screening Genetic risk of breast cancer

BRCA1 and BRCA2 mutation carriers have a significant cumulative lifetime risk of developing breast cancer, estimated to be 65% and 45%, respectively by the age of 70 [42]. NICE guidelines recommend that these high risk women receive annual MRI screening from the age of 30, with the addition of annual XRM from the age of 40. At 50, continuation of MRI screening is dependent on breast density [43][44]. The Royal Marsden NHS Foundation Trust screened a large number of these women until 2013, when they were repatriated back into the NHS Breast Screening Service. At St George's Hospital NHS Trust, screening is currently taking place as a part of the NHS Breast Screening Service. Investigators will retrospectively analyse MRI and XRM examinations from women who were aged between 40 and 50 years at screening.

Cohort 3: Participants attending MRI & XRM for breast screening post mantle radiotherapy Environmental risk of breast cancer

Treatment with high dose mantle radiotherapy at a young age also confers a much higher risk of breast cancer than that of the general population, estimated to result in an increased relative risk of 14.4 in comparison with the general population. NICE guidelines recommend that these high risk women receive annual MRI screening from the age of 30, with the addition of annual XRM from the age of 40. At 50, continuation of MRI screening is dependent on breast density. The Royal Marsden NHS Foundation Trust screened a large number of these women until 2013, when they were repatriated back into the NHS Breast Screening Service. At St George's Hospital NHS Trust, screening is currently taking place as a part of the NHS Breast Screening Service. Investigators will retrospectively analyse MRI and XRM examinations from women who were aged between 40 and 50 years at screening.

Cohort 4: General population attending XRM for breast investigation Population risk of breast cancer

Symptomatic women within the general population are referred to the Rapid Diagnostic and Assessment Centre (RDAC) for breast investigations. A series of diagnostic tests are performed at the RDAC which can include XRM if the women are 40 years of age or above. MRI is not normally performed in this setting. Significant numbers of these women are found to have normal breast tissue at XRM. These are women who have a population (low) risk of breast cancer but who might potentially benefit from an MRI investigation. Investigators will prospectively invite these women for a clinical MRI breast screening examination.

The aim of this study is to develop quantitative MRI measurements of breast tissue from clinical MRI breast protocols and to demonstrate that these descriptors have potential value for breast cancer risk prediction.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

* Normal breast tissue in one or both breasts
* Aged > 39.5 years
* ≤ 6 months between XRM and MRI examinations

Cohort 2:

* Genetically proven BRCA1 or 2 mutation carrier
* Age 39.5 - 50.5 years
* ≤ 6 months between XRM and MRI examinations

Cohort 3:

* Previous mantle radiotherapy
* Age 39.5 - 50.5 years
* ≤ 6 months between XRM and MRI examinations

Cohort 4:

* Radiologically healthy breast tissue as assessed by XRM
* Age 39.5 - 50.5 years
* Able to attend MRI screening within 6 weeks of XRM

Exclusion Criteria:

Cohort 1:

- Treatment or medication between XRM and MRI examinations

Cohort 2:

* Previous breast cancer diagnosis and/or treatment
* Treatment or medication between XRM and MRI examinations

Cohort 3:

* Previous breast cancer diagnosis and/or treatment
* Treatment or medication between XRM and MRI examinations

Cohort 4:

* Previous breast cancer diagnosis and/or treatment
* MRI incompatible implants
* Claustrophobia
* Inability to tolerate a 40 minute MRI breast examination
* Patients with renal failure or problems with IV access

Ages: 39 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Cohort 1:
  Retrospective breast MRI and XRM exam from participants with a clinical indication, reported as normal.
  Cohort 2:
  Retrospective breast MRI and XRM exams from genetically-proven BRCA1 or BRCA2 carriers; attendance at High Risk Breast Screening Service, RMH, and St George's Hospital (SGH).
  Cohort 3:
  Retrospective breast MRI and XRM exams from participants who received mantle radiotherapy at a young age and who subsequently attended the historic High Risk Breast Screening Service at RMH, or the High Risk Breast Screening Service at SGH.
  Cohort 4:
  Participants attending the RMH Rapid Diagnostic Assessment Centre for breast investigations who are found to have normal breast tissue on XRM will be prospectively invited for a breast MRI exam with administration of contrast agent.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Arm 1 (Cohort 1), Arm 2 (Cohorts 2 & 3) : breast density | After retrospective selection of subject groups (approximately 6 months).
  Breast density is measured in standard clinical sequences and in research sequences, expected to be the gold standard, as a %volume.
Arm 1 (Cohort 1), Arm 2 (Cohorts 2-3) : breast parenchyma enhancement (BPE) | After retrospective selection of subject groups (approximately 6 months).
  BPE is measured as a % of pre-contrast image intensity on dynamic contrast-enhanced examinations.
Arm 2 (Cohort 4): breast density | Six months after recruitment
  Breast density is measured in standard clinical sequences and in research sequences, expected to be the gold standard, as a %volume.
Arm 2 (Cohort 4): breast parenchyma enhancement (BPE) | Six months after recruitment
  BPE is measured as a % of pre-contrast image intensity on dynamic contrast-enhanced examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Allen, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom